CLINICAL TRIAL: NCT03711890
Title: Imaging and Detection of Micrometer Sized Early Stage Pancreatic Cancer by Using Endoscopic Ultra-High Resolution Optical Coherence Tomography (OCT) Using Resected Pancreatic Specimen, a Pilot Study
Brief Title: Ultra-High Resolution Optical Coherence Tomography in Detecting Micrometer Sized Early Stage Pancreatic Cancer in Participants With Pancreatic Cancer
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Mary Dillhoff, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-18060; NCI-2018-01534 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-08-13; First posted 2018-10-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Carcinoma; Pancreatic Intraductal Papillary Mucinous Neoplasm, Pancreatobiliary-Type
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Intraductal Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (resection, OCT) (Experimental): Participants undergo resection. Resected tissues are analyzed via ultra-high resolution OCT.
  Interventions: Procedure: Optical Coherence Tomography; Procedure: Therapeutic Conventional Surgery; Diagnostic Test: Laboratory Evaluation

INTERVENTIONS:
Procedure: Optical Coherence Tomography — Undergo OCT
  Other Names: OCT
Procedure: Therapeutic Conventional Surgery — Undergo resection will be undertaken
Diagnostic Test: Laboratory Evaluation — Labs will be obtained to test for cancer cell derived exosomes

SUMMARY:
This trial studies how well ultra-high resolution optical coherence tomography works in detecting micrometer sized early stage pancreatic cancer in participants with pancreatic cancer. Ultra-high resolution optical coherence tomography may help to accurately identify pancreatic cancer in resected pancreatic specimens.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the using of optical coherence tomography (OCT) to diagnose pancreatic cancer arising in the setting of intraductal papillary mucinous neoplasms (IPMN) using the resected pancreatic specimen.

II. To correlate OCT imaging diagnosis with histologic findings in the human pancreatic duct.

IPMN is a premalignant lesions arising in the pancreas. Typically, IPMNs are identified incidentally on imaging performed for other reason or related to vague abdominal pain or gastrointestinal complaints. In terms of IPMN, invasive cancer can be found in this setting between 20 to 50% of the time[7] Therefore, if a patient is diagnosed with IPMN, especially main duct type, the general recommendation is to undergo resection. We propose to assess the duct of the pancreatic specimen after resection to identify evidence of invasive malignancy by OCT imaging. Afterwards, the specimen will be undergoing histopathologic assessment using standard protocols. Our hypothesis is that OCT will accurately identify pancreatic cancer in resected pancreatic specimen. The assessment with OCT is non-invasive and will not harm to change the specimen prior to going to pathology for standard review. Future studies will then focus on using this imaging technique in vivo to endoscopically identify early stage pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Immediate surgery cohort: Adult patients with pancreatic cancer or IPMN
* Immediate surgery cohort: Informed consent will be obtained
* Adult patients undergoing pancreatic resection for a presumed IPMN

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure accuracy of using OCT to diagnose pancreatic cancer and compare with histology. | Up to 3 years
  Will evaluate the accuracy of the optical coherence tomography (OCT) based diagnosis compare to the pathological diagnosis or the cancer cell derived exosomes test from the blood sample. Will compare the diagnosis results from the OCT imaging technology to standard histopathologic assessment and the blood test using 2-way tables. The agreement between two tests will be summarized with the overall agreement and the Cohen?s Kappa values.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dillhoff, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamelinesline — http://cancer.osu.edu